CLINICAL TRIAL: NCT06783673
Title: Clinicopathological, Endoscopic and Serological Patterns of Celiac Disease in Children at Sohag University Hospital
Brief Title: Celiac Disease in Children
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Ali Abdelraheem, pediatrician, Sohag University
Other Study IDs: Soh-Med--24-11-10MS
Record Dates: First submitted 2024-12-30; First posted 2025-01-20 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Celiac Disease in Children
Keywords: clinicopathological, endoscopic and serological patterns of celiac disease in children
MeSH Terms: interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patterns of celiac disease in children: clinicopathological, endoscopic and serological patterns of celiac disease in children
  Interventions: Procedure: Upper GIT endoscopy

INTERVENTIONS:
Procedure: Upper GIT endoscopy — upper GIT endoscopy of suspected cases and multiple biopsies will be taken for histopathological examination
  Other Names: Upper endoscopy

SUMMARY:
The aim is to study the clinical, serological, endoscopic and histopathological characteristics and treatment outcome of children diagnosed with celiac disease in Sohag University Hospital

DETAILED DESCRIPTION:
Celiac disease (CD), or gluten-sensitive enteropathy, is an immune-mediated enteropathy triggered by the ingestion of gluten-containing cereals (wheat, barley, and rye) in genetically susceptible individuals. Undiagnosed CD may cause intestinal (e.g. chronic diarrhea, failure to thrive) and/or extra intestinal (e.g. anemia, osteoporosis, dermatitis herpetiformis) manifestations.

The etiology of CD is multifactorial, with both genetic and environmental factors involved in disease development. Susceptibility to CD is primarily associated with the human leukocyte antigen HLA-DQ2 allele. The heterodimer DQA1*0501 and DQB1*0201 is detected in up to 95% of persons with celiac disease, with the remaining 5% expressing HLA-DQ8 (DQA1*0301, DQB1*0302). The frequency of these alleles in the general populations in Western countries is 20% to 30%. Therefore, an individual not carrying DQ2 or DQ8 alleles is extremely unlikely to develop CD.

Celiac disease is associated with a host of autoimmune diseases such as type 1 diabetes mellitus, autoimmune thyroid disease, Addison disease, autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, and immunoglobulin (Ig) A deficiency. There is also an increased prevalence of CD in patients with genetic disorders such as Down syndrome and Turner syndrome.

Serologic testing is recommended as the first step in pursuing a diagnosis of CD, however, small-bowel mucosal biopsy is currently considered the gold standard for diagnosing CD. All serologic tests and small-bowel biopsies need to be performed while the patient is on a gluten-containing diet.

The characteristics of small intestine biopsies from CD include partial or complete villous atrophy, crypt hyperplasia, and intraepithelial lymphocyte infiltration.

According to the modified Marsh classification, the intestinal damage is divided into four stages. Stage 0 intestinal damage is characterized by the lesion invasion in the mucous layer, the increased number of intraepithelial lymphocytes and the presence of lymphocytes in the lamina propria, whereas Stage 1 damage features microscopic enteritis with an increase of intraepithelial lymphocytes. A feature of Stage 2 intestinal damage is crypt hyperplasia along with villous atrophy while Stage 3 is characterized by a complete atrophy of the intestinal villi.

Treatment of CD includes lifelong gluten-free diet. The clinical and histological benefits of a gluten-free diet (GFD) in the management of CD are well recognized showing that the degree of histological recovery is dependent upon how strict the patient adheres to the diet.

ELIGIBILITY:
Inclusion Criteria:

* Children less than 18 years.
* Both sexes.
* Children suffering from manifestations of celiac disease.
* Children previously diagnosed with celiac disease.

Exclusion Criteria:

* cases more than 18 years.
* Children diagnosed with other causes of malabsorption

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will include children who will be admitted to the department of pediatrics at Sohag University Hospital during the study period and which will be fulfilling the following eligibility criteria in addition to all children previously diagnosed with celiac disease in the last 1 years.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2024-08-25 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with Clinicopathological, endoscopic and serological patterns of Celiac disease | 1 Year
  clinical patterns of celiac disease include intestinal and extraintestinal manifestations.
  serological patterns include total IgA level, tissue transglutaminase IgA & IgG levels and endomesial IgA & IgG levels.
  Endoscopic patterns include patchy or generalized atrophy and scalloping of duodenal mucosa.
  Pathological patterns include features of mucosal atrophy and modified Marsh classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided